CLINICAL TRIAL: NCT00222352
Title: Diagnosis and Treatment of Acute Coronary Syndromes in the Emergency Department: The Impact of Rapid Bedside cTnI Testing on Outcomes
Brief Title: Diagnosis and Treatment of ACS in the ED: The Impact of Rapid Bedside cTnI Testing on Outcomes
Acronym: Dispo-ACS
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: Abbott (Industry); Jewish Hospital, Cincinnati, Ohio (Other); University of Pennsylvania (Other); Stanford University (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian Gibler, Study Chairman, University of Cincinnati
Other Study IDs: TJH 04-28
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Angina, Unstable
Keywords: Unstable Angina; Non-ST-segment Myocardial Infarction; Myocardial Necrosis; Troponin I
MeSH Terms: conditions — Angina, Unstable; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — SERUM BANKING Each patient consented and enrolled will have whole blood and plasma saved and frozen. The amount of blood drawn for the study is 5 ml (per draw), which is to be placed in a lithium heparinzed tube. One ml of whole blood will be alloquoted, frozen at -70ºC, and shipped to the Study Coordinating Center. The remainder of the sample will be centrifuged, alloquoted, frozen at -70ºC, and shipped to the Study Coordinating Center. These blood samples will be de-identified and assigned a study ID #. There will be no genetic testing of these samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- central laboratory cTnI test: Control Group
- Point of Care cTnL testing: Experimental Group
  Interventions: Diagnostic Test: Point of Care cTnL testing

INTERVENTIONS:
Diagnostic Test: Point of Care cTnL testing — The study design will be a phase IV prospective, randomized (1:1), parallel-group trial utilizing concurrent controls. The experimental group of interest will be patients receiving the POC cTnI test, and the control group will be patients receiving the central laboratory cTnI test.
  The treating physician will be blinded to the randomization and will receive only the POC results from half the study patients and only the laboratory results for the remaining half.
  Groups: Point of Care cTnL testing

SUMMARY:
In a randomized, controlled clinical trial, point-of care testing at the bedside using the cardiac biomarker troponin I in ED patients with possible ACS will be compared to traditional testing of this assay for myocardial necrosis obtained in the central laboratory. Our hypothesis: point-of-care testing for troponin I will decrease the time for disposition of patients with possible ACS in the emergency setting and decrease the time required for administering appropriate therapies for these patients.

DETAILED DESCRIPTION:
Cardiac troponin I is routinely used in the emergency department as a risk stratification tool for detecting myocardial necrosis in patients with possible acute coronary syndrome. It is our hypothesis that having bedside, point-of-care testing for TnI in the ED will decrease time needed to disposition patients to home from the ED or send to the cardiac catheterization laboratory or intensive care setting. Similarly, having point-of-care testing in the ED should decrease the time required to deliver anti-platelet drugs such as aspirin and glycoprotein IIb/IIIa inhibitors and anti-thrombin agents such as heparin to high risk patients found to have a positive TnI test. This will be evaluated in a randomized, controlled clinical trial of 2000 patients. Half will have the test performed in the ED at the bedside (point-of-care) while the other half will receive the usual lab results obtained from the central lab (typically requiring 1.5-2 hours to return).

ELIGIBILITY:
Inclusion criteria

* Age >21 years old
* Chest pain or other symptoms that lead to drawing cardiac bio-markers for possible ACS diagnosis

Exclusion criteria

* Presentation with chest pain in the presence of a tachydysrhythmia (ventricular tachycardia, supraventricular tachycardia, or rapid atrial fibrillation)
* Presentation with ECG diagnostic for STEMI

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 21 years or older, presenting with symptoms suggestive of acute coronary syndromes, and having cardiac biomarker tests ordered by the treating emergency physician were enrolled. Patients with a tachydysrhythmia (ventricular tachycardia, supraventricular tachycardia, or rapid atrial fibrillation) or a 12-lead ECG diagnostic for acute myocardial infarction were excluded. Patients were enrolled at 4 sites across the United States between December 2004 and November 2006, with final data collection and verification occurring by March 2007.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2006-11 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Time to disposition from the ED | The time from blood draw to initiation of therapy or to disposition
  The primary hypotheses are that i) POC testing using the i-STAT system reduces the time to disposition and discharge for low-risk patients being discharged directly from the ED, and ii) POC testing using the i-STAT system reduces the time to therapy compared to laboratory testing for the subset of patients requiring anti-thrombotic therapies such as heparin/LMW heparin or anti-platelet agents such as GPIIb/IIIa inhibitors or clopidogrel or PCI. These groups of patients (those with new ST-depression, recurrent pain, positive troponin, diabetes, age >65 years, or failed ASA and those discharged without a diagnosis associated with ischemic chest pain) will be extracted from the entire sample. The time from blood draw to initiation of therapy or to disposition and discharge will be computed and compared between the group with POC testing and the group with laboratory testing.

SECONDARY OUTCOMES:
Time to departure | time of discharge to home or to the time of transfer to an inpatient setting

CONTACTS AND LOCATIONS:
Overall Officials: Walter B Gibler, MD, Study Chair — University of Cincinnati
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - William Beaumont Hospital, Royal Oak, Michigan
  - The Jewish Hospital, Cincinnati, Ohio
  - The University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
Blood samples banked for future use. Must be IRB approved before use.